CLINICAL TRIAL: NCT06334731
Title: What Happened? Antimicrobial Resistance During the SARS-CoV-2 (COVID-19) Pandemic
Brief Title: Antimicrobial Resistance During the SARS-CoV-2 (COVID-19) Pandemic
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 045.PHA.2021.D
Record Dates: First submitted 2022-10-21; First posted 2024-03-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Assess the incidence and rates of resistant pathogens prior to and during the COVID-19 pandemic.

DETAILED DESCRIPTION:
The COVID-19 pandemic accelerated/exacerbated resistance rates for key pathogens. Specifically, incidence of extended-spectrum beta-lactamase producing Enterobacteriaceae (ESBLPE), carbapenem-resistant bacteria (CRB), methicillin-resistant Staphyloccoccus aureus (MRSA), vancomycin-resistant Enterococci (VRE), and C. difficile infections (CDI) will be higher in the pandemic time period (Pandemic, March 2020 - February 2025) compared to the pre-pandemic period (Pre-Pandemic, March 2018 - February 2020).

ELIGIBILITY:
Inclusion Criteria:

* • Patients admitted to Methodist Richardson, Methodist Mansfield, Methodist Charlton, or Methodist Dallas Medical Centers between March 2018 and August 2021.

  * >18 years old

Exclusion Criteria:

* • Outpatient visit

  * Not admitted to an inpatient or observation status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Methodist Richardson, Methodist Mansfield, Methodist Charlton, or Methodist Dallas Medical Centers between March 2018 and August 2021.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Incidence of third generation cephalosporin-resistant bacteria (3GCRB) | 5 Months
  Incidence of third generation cephalosporin-resistant bacteria (3GCRB)

SECONDARY OUTCOMES:
Incidence of ESBLPE | 5 months
  Incidence of ESBLPE
Incidence of CRB | 5 Months
  Incidence of CRB
Incidence of other pathogens | August 2021
  * MRSA
  * VRE
  * CDI
Incidence of nosocomial infections | 5 Months
  * Catheter-associated urinary tract infection (CAUTI)
  * Central line-associated bloodstream infection (CLABSI)
  * Possible ventilator-associated pneumonia (PVAP)
Incidence of clinical outcomes | 5 Months
  death, recovery, long-term care facility, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Crotty, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No